CLINICAL TRIAL: NCT05094934
Title: Investigation of Pharmacokinetics, Safety and Tolerability of Oral NNC0385-0434 in Participants With Various Degrees of Impaired Renal Function and in Participants With Normal Renal Function
Brief Title: A Research Study Looking Into Levels of the Medicine NNC0385-0434 in the Body and How Well it is Tolerated in Participants With Impaired Kidney Function Compared to Participants With Normal Kidney Function
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN6435-4749; U1111-1264-2693 (Other: World Health Organization (WHO)); 2021-000462-16 (EudraCT Number)
Record Dates: First submitted 2021-09-27; First posted 2021-10-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal renal function (Active Comparator): All participants will receive 100 mg of NNC0385-0434 in an oral tablet per day for 10 days
  Interventions: Drug: NNC0385-0434 A 100 mg
- Mildly decreased renal function (Experimental): All participants will receive 100 mg of NNC0385-0434 in an oral tablet per day for 10 days
  Interventions: Drug: NNC0385-0434 A 100 mg
- Moderately decreased renal function (Experimental): All participants will receive 100 mg of NNC0385-0434 in an oral tablet per day for 10 days
  Interventions: Drug: NNC0385-0434 A 100 mg
- Severely decreased renal function (Experimental): All participants will receive 100 mg of NNC0385-0434 in an oral tablet per day for 10 days
  Interventions: Drug: NNC0385-0434 A 100 mg

INTERVENTIONS:
Drug: NNC0385-0434 A 100 mg — All participants will receive the same dose (100 mg) of the study medicine NNC0385-0434, which will be given for 10 days in a row. Participants will get the study medicine in a tablet taken orally once-daily. The study medicine needs to be taken in the morning after overnight fasting and 30 minutes before the first meal of the day.

SUMMARY:
Novo Nordisk is developing a new medicine, NNC0385-0434, to help people lower their cholesterol level.

The aim of this study is to look at how NNC0385-0434 works in the body and how it is removed from the body in people with impaired kidney function.

All participants will receive the same dose (100 mg) of the study medicine NNC0385-0434, which will be given for 10 days in a row. Participants will get the study medicine in a tablet taken orally once-daily. The study medicine needs to be taken in the morning after overnight fasting and 30 minutes before the first meal of the day.

The study will last for about 9-14 weeks.

Participants will have 15 visits to the study centre, including 2 in-house stays of 3 days and 2 nights and 13 ambulatory visits.

Participants' vital signs (heart rate, blood pressure, body temperature) will be measured, participants will have blood draws, urine will be collected and electrocardiograms (ECGs) will be recorded.

Participants cannot take part in the study if they have gastrointestinal disorders or unusual meal habits and special dietary requirements.

Women can only take part in the study if they cannot get pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 20.0 and 34.9 kg/m^2 (both inclusive).
* Meeting the pre-defined estimated glomerular filtration rate (eGFR) values based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation according to KDIGO 2012:

Group description eGFR (mL/min)

1. Normal renal function more than or equal to 90
2. Mildly decreased renal function 60 - less than 90
3. Moderately decreased renal function 30 - less than 60
4. Severely decreased renal function less than 30 not requiring dialysis

Exclusion Criteria:

* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the study doctor.
* Unusual meal habits and special dietary requirements or unwillingness to eat the food provided in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,0434,Day10: the area under the NNC0385-0434 plasma concentration-time curve from time 0 to 24 hours after last dose of oral NNC0385-0434 | From last dose (Day 10) to 24 hours post treatment (Day 11)
  Measured in h*nmol/L

SECONDARY OUTCOMES:
Cmax,0434,Day10: the maximum plasma concentration of NNC0385-0434 after last dose of oral NNC0385-0434 | From last dose (Day 10) to post treatment follow-up (Day 65)
  nmol/L
tmax,0434,Day10: time from last dose administration to maximum plasma concentration of oral NNC0385-0434 | From last dose (Day 10) to post treatment follow-up (Day 65)
  h
t½,0434,Day10; the terminal half-life of NNC0385-0434 after last dose of oral NNC0385-0434 | From last dose (Day 10) to post treatment follow-up (Day 65)
  h
CLR,0434,Day10; the renal clearance of NNC0385-0434 after last dose of oral NNC0385-0434 | From last dose (Day 10) to 48 hours post treatment (Day 12)
  mL/h
AUC0-24h,SNAC,Day10: the area under the SNAC plasma concentration-time curve from time 0 to 24 hours after last dose of oral NNC0385-0434 | From last dose (Day 10) to 24 hours post treatment (Day 11)
  h*ng/mL
Cmax,SNAC,Day10; the maximum plasma concentration of SNAC after last dose of oral NNC0385-0434 | From last dose (Day 10) to 24 hours post treatment (Day 11)
  ng/mL
Cmin,SNAC,Day10; the minimum plasma concentration of SNAC before last dose of oral NNC0385-0434 | Pre-dose (Day 10)
  nmol/L
tmax,SNAC,Day10; the time to maximum observed plasma concentration of SNAC after last dose of oral NNC0385-0434 | From last dose (Day 10) to 24 hours post treatment (Day 11)
  hours
CLR,SNAC,Day10; the renal clearance of SNAC after last dose of oral NNC0385-0434 | From last dose (Day 10) to 48 hours post treatment (Day 12)
  mL/h
Number of treatment emergent adverse events (TEAEs) | From first dose (Day 1) until completion of the post-treatment period at follow-up (Day 65)
  Number of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com